CLINICAL TRIAL: NCT06109233
Title: A Perspective Study of the MRD-tailored Therapy in Patients With Newly Diagnosed Multiple Myeloma With Persistent Minimal Residual Disease After Initial Treatment
Acronym: MRD
Status: Recruiting | Type: Observational
Sponsor: FengYan Jin (Other)
Responsible Party: Sponsor-Investigator, FengYan Jin, Clinical Professor of Hematology Department, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: MRD 2023
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Minimal Residual Disease
Keywords: Multiple Myeloma; MRD-tailored therapy; MRD status; MRD-negative rates; Survival
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood、bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRD negativity: NDMM patients who obtained MRD negativity after induction and consolidation therapy
- MRD positivity: NDMM patients who MRD positivity after induction and consolidation therapy and agree to adjust the treatment regimen

SUMMARY:
The aim of this study was to observe the rate of MRD conversion and the impact on survival in newly diagnosed multiple myeloma (NDMM) patients with persistent MRD positivity after induction and consolidation therapy (autologous hematopoietic stem cell transplantation or consolidation of the original regimen) who were switched to high-intensity therapy, and to compare the rate of persistent MRD-negativity, progression-free survival (PFS), and overall survival (OS) between the two groups in comparison with NDMM patients who achieved MRD-negativity after the same induction and consolidation therapy.

DETAILED DESCRIPTION:
There is still an unmet clinical need as to whether NDMM patients with persistent MRD positive would benefit from switching to high-intensity therapy. The induction regimen (Dara+/- (Vd, Rd, Pd, VRd, VPd)) was selected based on the frail or high-risk status of NDMM patients. Transplantation or consolidation and maintenance regimens were adjusted by MRD status detected by NGF.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have documented newly diagnosed symptomatic multiple myeloma as defined by 2014 International Myeloma Working Group criteria.
3. Subject must have achieved a response (partial response [PR] or better based on investigator's determination of response by the IMWG criteria) to at one prior regimen.
4. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. Contraception must begin 4 weeks prior to dosing and continue until at least 3 months after receiving the last dose of the study drug. A woman of childbearing potential must have a negative serum or urine pregnancy tests at screening within 14 days prior to randomization.
5. Each subject (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma. Monoclonal gammopathy of undetermined significance is defined by presence of serum M-protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the M-protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less. Smoldering multiple myeloma is defined as asymptomatic multiple myeloma with absence of related organ or tissue impairment or end-organ damage.
2. Relapsed and refractory myeloma：Relapsed and refractory myeloma is defined as disease that is nonresponsive while on salvage therapy, or progresses within 60 days of last therapy in patients who have achieved minimal response (MR) or better at some point previously before then progressing in their disease course.
3. Primary refractory myeloma：Primary refractory myeloma is defined as disease that is nonresponsive in patients who have never achieved a minimal response or better with any therapy.
4. Subject is known or suspected of not being able to comply with the study protocol。 Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with multiple myeloma according to the 2014 IMWG multiple myeloma diagnostic criteria, receiving induction and consolidation therapy to achieve partial remission (PR) or better, and MRD-negative, or persistently MRD-positive and agreeing to adjust the treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Adjusted treatment-adjusted MRD-negative rates | through study completion, up to 2 years
  To explore the rate of conversion to MRD-negative after adjusting treatment in NDMM patients with persistent MRD-positive status.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, up to 2 years
  PFS were calculated from the enrollment to the first instance of disease progression, relapse, or death
Overall Survival (OS) | through study completion, up to 2 years
  OS were calculated from the time of enrollment to death or the last follow-up
Persistent MRD-negative rates and survival | through study completion, up to 2 years
  Persistent MRD-negative rates and survival (including PFS and OS) in both groups compared to NDMM patients who achieved MRD-negativity after the same induction and consolidation therapy
Treatment related adverse event(TRAE) | through study completion, up to 2 years
  Toxicity and safety will be reported based on the adverse events, as graded by CTCAE V5 and determined by routine clinical assessments.

OTHER OUTCOMES:
explore the molecular basis for the dynamic changes and differences in MRD | through study completion, up to 2 years
  Bone puncture samples from routine clinical consultations were collected, and single-cell transcriptome sequencing technology was applied to analyze and compare the differences in MM cells (clones) and bone marrow microenvironment (including immunity, inflammation, and stroma) of MRD-transformed and non-transformed patients after adjusting the treatment regimen, using the samples before adjusting the treatment regimen as the baseline control, in order to explore the molecular basis for the dynamic changes and differences in MRD
explore the elderly (especially debilitated) patients' MRD-adjusted treatment | through study completion, up to 2 years
  For patients ≥65 years old, through the adjusted treatment-adjusted MRD-negative rates to explore the impact of strategy adjustment on elderly patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar SK, Rajkumar V, Kyle RA, van Duin M, Sonneveld P, Mateos MV, Gay F, Anderson KC. Multiple myeloma. Nat Rev Dis Primers. 2017 Jul 20;3:17046. doi: 10.1038/nrdp.2017.46. PMID 28726797
- [Background] Anderson KC. Progress and Paradigms in Multiple Myeloma. Clin Cancer Res. 2016 Nov 15;22(22):5419-5427. doi: 10.1158/1078-0432.CCR-16-0625. PMID 28151709
- [Background] Kumar SK, Rajkumar SV. The multiple myelomas - current concepts in cytogenetic classification and therapy. Nat Rev Clin Oncol. 2018 Jul;15(7):409-421. doi: 10.1038/s41571-018-0018-y. PMID 29686421
- [Background] Maiso P, Huynh D, Moschetta M, Sacco A, Aljawai Y, Mishima Y, Asara JM, Roccaro AM, Kimmelman AC, Ghobrial IM. Metabolic signature identifies novel targets for drug resistance in multiple myeloma. Cancer Res. 2015 May 15;75(10):2071-82. doi: 10.1158/0008-5472.CAN-14-3400. Epub 2015 Mar 13. PMID 25769724
- [Background] Alonso S, Hernandez D, Chang YT, Gocke CB, McCray M, Varadhan R, Matsui WH, Jones RJ, Ghiaur G. Hedgehog and retinoid signaling alters multiple myeloma microenvironment and generates bortezomib resistance. J Clin Invest. 2016 Dec 1;126(12):4460-4468. doi: 10.1172/JCI88152. Epub 2016 Oct 24. PMID 27775549
- [Background] Paiva B, Puig N, Cedena MT, de Jong BG, Ruiz Y, Rapado I, Martinez-Lopez J, Cordon L, Alignani D, Delgado JA, van Zelm MC, Van Dongen JJ, Pascual M, Agirre X, Prosper F, Martin-Subero JI, Vidriales MB, Gutierrez NC, Hernandez MT, Oriol A, Echeveste MA, Gonzalez Y, Johnson SK, Epstein J, Barlogie B, Morgan GJ, Orfao A, Blade J, Mateos MV, Lahuerta JJ, San-Miguel JF. Differentiation stage of myeloma plasma cells: biological and clinical significance. Leukemia. 2017 Feb;31(2):382-392. doi: 10.1038/leu.2016.211. Epub 2016 Aug 1. PMID 27479184
- [Background] Jelinek T, Bezdekova R, Zatopkova M, Burgos L, Simicek M, Sevcikova T, Paiva B, Hajek R. Current applications of multiparameter flow cytometry in plasma cell disorders. Blood Cancer J. 2017 Oct 20;7(10):e617. doi: 10.1038/bcj.2017.90. PMID 29053157
- [Background] Flores-Montero J, Sanoja-Flores L, Paiva B, Puig N, Garcia-Sanchez O, Bottcher S, van der Velden VHJ, Perez-Moran JJ, Vidriales MB, Garcia-Sanz R, Jimenez C, Gonzalez M, Martinez-Lopez J, Corral-Mateos A, Grigore GE, Fluxa R, Pontes R, Caetano J, Sedek L, Del Canizo MC, Blade J, Lahuerta JJ, Aguilar C, Barez A, Garcia-Mateo A, Labrador J, Leoz P, Aguilera-Sanz C, San-Miguel J, Mateos MV, Durie B, van Dongen JJM, Orfao A. Next Generation Flow for highly sensitive and standardized detection of minimal residual disease in multiple myeloma. Leukemia. 2017 Oct;31(10):2094-2103. doi: 10.1038/leu.2017.29. Epub 2017 Jan 20. PMID 28104919
- [Background] Puig N, Sarasquete ME, Balanzategui A, Martinez J, Paiva B, Garcia H, Fumero S, Jimenez C, Alcoceba M, Chillon MC, Sebastian E, Marin L, Montalban MA, Mateos MV, Oriol A, Palomera L, de la Rubia J, Vidriales MB, Blade J, Lahuerta JJ, Gonzalez M, Miguel JF, Garcia-Sanz R. Critical evaluation of ASO RQ-PCR for minimal residual disease evaluation in multiple myeloma. A comparative analysis with flow cytometry. Leukemia. 2014 Feb;28(2):391-7. doi: 10.1038/leu.2013.217. Epub 2013 Jul 17. PMID 23860448
- [Background] Silvennoinen R, Lundan T, Kairisto V, Pelliniemi TT, Putkonen M, Anttila P, Huotari V, Mantymaa P, Siitonen S, Uotila L, Penttila TL, Juvonen V, Selander T, Remes K. Comparative analysis of minimal residual disease detection by multiparameter flow cytometry and enhanced ASO RQ-PCR in multiple myeloma. Blood Cancer J. 2014 Oct 10;4(10):e250. doi: 10.1038/bcj.2014.69. PMID 25303369
- [Background] Martinez-Lopez J, Lahuerta JJ, Pepin F, Gonzalez M, Barrio S, Ayala R, Puig N, Montalban MA, Paiva B, Weng L, Jimenez C, Sopena M, Moorhead M, Cedena T, Rapado I, Mateos MV, Rosinol L, Oriol A, Blanchard MJ, Martinez R, Blade J, San Miguel J, Faham M, Garcia-Sanz R. Prognostic value of deep sequencing method for minimal residual disease detection in multiple myeloma. Blood. 2014 May 15;123(20):3073-9. doi: 10.1182/blood-2014-01-550020. Epub 2014 Mar 19. PMID 24646471
- [Background] Avet-Loiseau H. Minimal Residual Disease by Next-Generation Sequencing: Pros and Cons. Am Soc Clin Oncol Educ Book. 2016;35:e425-30. doi: 10.1200/EDBK_159088. PMID 27249750
- [Background] Perrot A, Lauwers-Cances V, Corre J, Robillard N, Hulin C, Chretien ML, Dejoie T, Maheo S, Stoppa AM, Pegourie B, Karlin L, Garderet L, Arnulf B, Doyen C, Meuleman N, Royer B, Eveillard JR, Benboubker L, Dib M, Decaux O, Jaccard A, Belhadj K, Brechignac S, Kolb B, Fohrer C, Mohty M, Macro M, Richardson PG, Carlton V, Moorhead M, Willis T, Faham M, Anderson KC, Harousseau JL, Leleu X, Facon T, Moreau P, Attal M, Avet-Loiseau H, Munshi N. Minimal residual disease negativity using deep sequencing is a major prognostic factor in multiple myeloma. Blood. 2018 Dec 6;132(23):2456-2464. doi: 10.1182/blood-2018-06-858613. Epub 2018 Sep 24. PMID 30249784
- [Background] Davies FE, Forsyth PD, Rawstron AC, Owen RG, Pratt G, Evans PA, Richards SJ, Drayson M, Smith GM, Selby PJ, Child JA, Morgan GJ. The impact of attaining a minimal disease state after high-dose melphalan and autologous transplantation for multiple myeloma. Br J Haematol. 2001 Mar;112(3):814-9. doi: 10.1046/j.1365-2141.2001.02530.x. PMID 11260088
- [Background] Paiva B, Vidriales MB, Cervero J, Mateo G, Perez JJ, Montalban MA, Sureda A, Montejano L, Gutierrez NC, Garcia de Coca A, de Las Heras N, Mateos MV, Lopez-Berges MC, Garcia-Boyero R, Galende J, Hernandez J, Palomera L, Carrera D, Martinez R, de la Rubia J, Martin A, Blade J, Lahuerta JJ, Orfao A, San Miguel JF; GEM (Grupo Espanol de MM)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Groups. Multiparameter flow cytometric remission is the most relevant prognostic factor for multiple myeloma patients who undergo autologous stem cell transplantation. Blood. 2008 Nov 15;112(10):4017-23. doi: 10.1182/blood-2008-05-159624. Epub 2008 Jul 31. PMID 18669875
- [Background] Rawstron AC, Child JA, de Tute RM, Davies FE, Gregory WM, Bell SE, Szubert AJ, Navarro-Coy N, Drayson MT, Feyler S, Ross FM, Cook G, Jackson GH, Morgan GJ, Owen RG. Minimal residual disease assessed by multiparameter flow cytometry in multiple myeloma: impact on outcome in the Medical Research Council Myeloma IX Study. J Clin Oncol. 2013 Jul 10;31(20):2540-7. doi: 10.1200/JCO.2012.46.2119. Epub 2013 Jun 3. PMID 23733781
- [Background] Rawstron AC, Gregory WM, de Tute RM, Davies FE, Bell SE, Drayson MT, Cook G, Jackson GH, Morgan GJ, Child JA, Owen RG. Minimal residual disease in myeloma by flow cytometry: independent prediction of survival benefit per log reduction. Blood. 2015 Mar 19;125(12):1932-5. doi: 10.1182/blood-2014-07-590166. Epub 2015 Feb 2. PMID 25645353
- [Background] Paiva B, Cedena MT, Puig N, Arana P, Vidriales MB, Cordon L, Flores-Montero J, Gutierrez NC, Martin-Ramos ML, Martinez-Lopez J, Ocio EM, Hernandez MT, Teruel AI, Rosinol L, Echeveste MA, Martinez R, Gironella M, Oriol A, Cabrera C, Martin J, Bargay J, Encinas C, Gonzalez Y, Van Dongen JJ, Orfao A, Blade J, Mateos MV, Lahuerta JJ, San Miguel JF; Grupo Espanol de Mieloma/Programa para el Estudio de la Terapeutica en Hemopatias Malignas (GEM/PETHEMA) Cooperative Study Groups. Minimal residual disease monitoring and immune profiling in multiple myeloma in elderly patients. Blood. 2016 Jun 23;127(25):3165-74. doi: 10.1182/blood-2016-03-705319. Epub 2016 Apr 26. PMID 27118453
- [Background] Landgren O, Devlin S, Boulad M, Mailankody S. Role of MRD status in relation to clinical outcomes in newly diagnosed multiple myeloma patients: a meta-analysis. Bone Marrow Transplant. 2016 Dec;51(12):1565-1568. doi: 10.1038/bmt.2016.222. Epub 2016 Sep 5. PMID 27595280
- [Background] Lahuerta JJ, Paiva B, Vidriales MB, Cordon L, Cedena MT, Puig N, Martinez-Lopez J, Rosinol L, Gutierrez NC, Martin-Ramos ML, Oriol A, Teruel AI, Echeveste MA, de Paz R, de Arriba F, Hernandez MT, Palomera L, Martinez R, Martin A, Alegre A, De la Rubia J, Orfao A, Mateos MV, Blade J, San-Miguel JF; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Depth of Response in Multiple Myeloma: A Pooled Analysis of Three PETHEMA/GEM Clinical Trials. J Clin Oncol. 2017 Sep 1;35(25):2900-2910. doi: 10.1200/JCO.2016.69.2517. Epub 2017 May 12. PMID 28498784
- [Background] Munshi NC, Avet-Loiseau H, Rawstron AC, Owen RG, Child JA, Thakurta A, Sherrington P, Samur MK, Georgieva A, Anderson KC, Gregory WM. Association of Minimal Residual Disease With Superior Survival Outcomes in Patients With Multiple Myeloma: A Meta-analysis. JAMA Oncol. 2017 Jan 1;3(1):28-35. doi: 10.1001/jamaoncol.2016.3160. PMID 27632282
- [Background] Harousseau JL, Avet-Loiseau H. Minimal Residual Disease Negativity Is a New End Point of Myeloma Therapy. J Clin Oncol. 2017 Sep 1;35(25):2863-2865. doi: 10.1200/JCO.2017.73.1331. Epub 2017 May 19. No abstract available. PMID 28525304
- [Background] Anderson KC. Should minimal residual disease negativity be the end point of myeloma therapy? Blood Adv. 2017 Mar 14;1(8):517-521. doi: 10.1182/bloodadvances.2016000117. eCollection 2017 Mar 14. PMID 29296970
- [Background] Sonneveld P. Should minimal residual disease negativity not be the end point of myeloma therapy? Blood Adv. 2017 Mar 14;1(8):522-525. doi: 10.1182/bloodadvances.2017000109. eCollection 2017 Mar 14. PMID 29296971
- [Background] Paiva B, van Dongen JJ, Orfao A. New criteria for response assessment: role of minimal residual disease in multiple myeloma. Blood. 2015 May 14;125(20):3059-68. doi: 10.1182/blood-2014-11-568907. Epub 2015 Apr 2. PMID 25838346
- [Background] Yang P, Xu W, Liang X, Yu S, Yi X, Liu M, Tian M, Yue T, Zhang Y, Yan Y, Hu Z, Guo Q, Zhang N, Wang J, Sun X, Hu R, Kumar SK, Dai Y, Jin F. Dynamic monitoring of minimal residual disease in newly-diagnosed multiple myeloma. Am J Hematol. 2023 Mar;98(3):E61-E64. doi: 10.1002/ajh.26810. Epub 2022 Dec 21. No abstract available. PMID 36540935